CLINICAL TRIAL: NCT04884243
Title: A Phase 2 Multicenter, Double-masked, Randomized, Vehicle-controlled, Parallel Study to Evaluate the Safety, Efficacy and Pharmacokinetics of CBT-006 in Patients With Meibomian Gland Dysfunction
Brief Title: Safety, Efficacy and Pharmacokinetics of CBT-006 in Patients With Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cloudbreak Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBT-CS102
Record Dates: First submitted 2021-05-05; First posted 2021-05-12 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-08

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CBT-006 (Placebo Comparator): Vehicle
  Interventions: Drug: CBT-006
- CBT-006 lower concentration (Experimental): lower concentration dose
  Interventions: Drug: CBT-006
- CBT-006 higher concentration (Experimental): higher concentration dose
  Interventions: Drug: CBT-006

INTERVENTIONS:
Drug: CBT-006 — ophthalmic solution
  Other Names: not apply

SUMMARY:
STUDY DESIGN

Structure:

Multicenter, randomized, double-masked, vehicle-controlled, parallel group study.

Duration:

3 months of TID treatment.

Treatment Groups, Dosing, and Treatment Regimen:

Study Treatment: CBT-006 topical ophthalmic solution Control Treatment: CBT-006 vehicle

DETAILED DESCRIPTION:
Structure:

Multicenter, randomized, double-masked, vehicle-controlled, parallel group study.

Duration:

3 months of TID treatment.

Treatment Groups, Dosing, and Treatment Regimen:

Study Treatment: CBT-006 topical ophthalmic solution Control Treatment: CBT-006 vehicle

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MGD in both eyes and meet the following:

  1. Ocular discomfort Score (ODS) ≥ 2
  2. Visual Analog Scale (VAS) level is 35-90% for at least 1 of the 7 categories
  3. Total Cornea staining grade ≥ 3
  4. Total meibum quality score (MQS) is between 6-17 from the sum of the 6 lower eyelid central glands in at least one lower eyelid
  5. TBUT ≤ 5 s
  6. Schirmer I Test (anaesthetized) ≥ 5 mm/5 min in study eye
  7. BCVA LogMAR ≥ +0.7 in each eye
* All patients of both genders ≥ 18 years
* Willing to withhold the use of artificial tears and lubricants during the treatment phase;
* Able to provide written informed consent and comply with study assessments for the full duration of the study.

Exclusion Criteria:

* Uncontrolled systemic disease in the opinion of the Investigator
* Active allergies with symptoms that may confound the data, active ocular infection requiring treatment, or ocular surface inflammatory disease unrelated to MGD or DED, including chalazion, inflamed pinguecula, and viral illness
* History of ocular herpes disease in either eye
* Incisional ocular surgery within 6 months or ocular laser surgery within 3 months
* Use of topical treatment of the eye/eyelid with antibiotics, NSAIDS, or vasoconstrictors to treat MGD or DED within 14 days of screening; steroids, cyclosporin A or lifitegrast within 28 days of screening
* Current or anticipated use of other topical ophthalmic medications in the study eye. (Patients must have discontinued the use of ophthalmic medications in the study eye for at least 2 weeks prior to the screening visit, the use of diagnostic medications as part of the eye exam prior to screening and artificial tears is allowed.)
* Anticipated wearing of contact lenses during any portion of the study. (Patients, who wear soft contact lenses should discontinue wearing them at least 3 days prior to screening visit. Patients wearing rigid gas permeable or hard contact lenses should discontinue wearing them at least 3 weeks prior to screening visit.)
* Active rosacea involving the eyelids within 60 days of screening
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days prior to entry into this study
* Any condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study
* Female patients who are pregnant, nursing, or planning a pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rong Yang, Study Director — Cloudbreak Therapeutics, LLC
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT-006 | CBT-006 Lower Concentration | CBT-006 Higher Concentration
Started | 32 | 30 | 30
Completed | 32 | 29 | 28
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-006 | CBT-006 Lower Concentration | CBT-006 Higher Concentration | Total
Number analyzed (Participants) | 32 | 30 | 30 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 24 | 61
  >=65 years | 13 | 12 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (6.98) | 61.3 (11.75) | 52.3 (13.23) | 58.6 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 12 | 50
  Male | 14 | 10 | 18 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 9 | 23
  Not Hispanic or Latino | 25 | 23 | 21 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 7 | 16
  White | 22 | 23 | 17 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 30 | 92
Intraocular Pressure of study eye related to safety [Mean (Standard Deviation); unit: mmHg] | 16.328 (2.1425) | 16.517 (2.5342) | 16 (2.6781) | 16.282 (0.21359)

OUTCOME MEASURES:

1. Primary Outcome: IOP of Study Eye Related to Safety
Description: Intraocular Pressure of study eye related to safety
Time Frame: 12 weeks
Population: Safety Population Study eye
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- CBT-006 Vehicle: Vehicle
  CBT-006: ophthalmic solution
Arm/Group | CBT-006 Vehicle | CBT-006 Lower Concentration | CBT-006 Higher Concentration
Number analyzed (Participants) | 32 | 30 | 30
mmHg | 16.547 (2.0882) | 16.328 (2.6230) | 16.241 (2.6647)

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | CBT-006 | CBT-006 Lower Concentration | CBT-006 Higher Concentration
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/32 | 3/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-006 (N=32) | CBT-006 Lower Concentration (N=30) | CBT-006 Higher Concentration (N=30)
ocular TEAEs (Eye disorders) | 1 (1) | 2 (2) | 2 (2)
Non-ocular TEAEs (General disorders) | 3 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04884243/Prot_SAP_000.pdf